CLINICAL TRIAL: NCT05800028
Title: Memory and Social Interactions: Study in Alzheimer's Disease and Semantic Progressive Aphasia
Brief Title: Memory and Social Interactions
Acronym: MEM&SO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Collaborators: University Hospital, Rouen (Other); Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A00198-35
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer Disease; Semantic Dementia
Keywords: Memory; Social Interaction; Personality; Alzheimer Disease; Aphasia, Primary Progressive
MeSH Terms: conditions — Alzheimer Disease; Frontotemporal Dementia; Aphasia, Primary Progressive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- AD group: 30 individuals aged between 50 and 85 years with probable Alzheimer's disease dementia with amnestic presentation and documented decline following the recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease.
  Interventions: Behavioral: Learning new information
- SPPA group: 16 individuals aged between 50 and 85 years with the semantic variant of primary progressive aphasia following the classification of primary progressive aphasia and its variants.
  Interventions: Behavioral: Learning new information
- HC group: 46 individuals without cognitive complain.
  Interventions: Behavioral: Learning new information
- Partners: 92 individuals without cognitive complaints. Each of these individuals will partner with one of the members of the experimental groups to carry out learning in social contexts.
  Interventions: Behavioral: Learning new information

INTERVENTIONS:
Behavioral: Learning new information — The purpose of this study is to test the effects of different social contexts when learning new information. Participants in the AD, SPPA, and HC experimental groups will be given tests to learn verbal information (location of drawings in a grid). The learning phases of these tests are presented in the form of a memory game in which participants are asked to make pairs of drawings by finding the second copy of the proposed pair by trial and error in a grid. After learning, a task of recognizing the position of the drawings in the grid is performed. Each participant will carry out this learning in three different conditions: 1) learning alone, 2) learning by observation of the reconstruction of the pairs of images by a partner, and 3) collaborative learning in which the two game partners discover and reconstruct the pairs together.

SUMMARY:
Memory and social interaction are intimately linked. On the one hand, social interaction is a privileged context for learning, and on the other hand, appropriate social interactions involve remembering the partners encountered and previous exchanges. People with Alzheimer's disease classic syndrome variant (AD) have a major impairment of episodic memory, while people with the semantic variant of primary progressive aphasia (SPPA) are characterized by semantic disorders in the foreground, associated with changes in their social behavior with a tendency to egocentricity. In both cases, patients frequently have reduced social interactions. Although social interaction situations seem to constitute a privileged learning context, their effectiveness for patients with cognitive disorders must be evaluated and the conditions under which they are effective must be established. The main objective of this study is to determine whether social interaction constitutes a beneficial context for learning new information and whether the presence of social behavior disorders alters this benefit. More broadly, the goal is to better understand the mechanisms underlying the possible beneficial effect of learning in social contexts and to clarify the links between memory performance in different social contexts, cognitive disorders, social behavioral changes and personality traits. Finally, a description will be made of the brain substrates associated with memory performance obtained during learning in social contexts in order to investigate their particularities. Thirty couples each including a person with AD, 16 couples each including a person with SPPA and 46 couples of persons without cognitive complaints (HC), one of which will be matched in gender and age to one of the patients, will be included in the study. Participants will perform image location learning in a grid, in three social contexts in which both members of the couple are involved: 1) simple presence of others, 2) by observation and 3) in collaboration. A psychometric assessment including social cognition and classical tests assessing memory, and questionnaires concerning global executive functioning, social behavior and personality will be offered to all participants. Patients in the AD and SPPA groups and the matched individual in the HC group will undergo anatomical and functional brain magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion criteria:

* AD group: Age between 50 and 85 years, Diagnosis of probable Alzheimer's disease dementia with amnestic presentation and documented decline following the recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease.
* SPPA group: Age between 50 and 85 years, Diagnosis of the semantic variant of primary progressive aphasia following the classification of primary progressive aphasia and its variants.
* HC group: Age between 50 and 85 years, Matched in age and sociocultural status with one of the AD or SPPA patients, No cognitive complain, No recent reduction in social or cognitive activities, No contraindication to MRI examination.
* Partners: Age over 18 years of age , No cognitive complaints, Social interactions of at least two hours per week for at least 5 years with one of the individuals of the other three groups.

Exclusion criteria (for all groups):

* Deprivation of liberty by judicial or administrative decision
* Not being a member of a social security system
* Concurrent participation in a therapeutic drug trial
* Uncorrected visual and/or auditory disorders that are sufficiently significant to interfere with the protocol
* History of neurological disorders (stroke, epilepsy, head trauma with loss of consciousness for more than one hour)
* History of chronic alcoholism or drug abuse
* History within the last 10 years of a clinically significant major psychiatric disorder
* Cancer within the past 5 years, except for squamous cell carcinoma
* Use of medications that may affect cognitive and/or brain function. Given the number of molecules involved and the dosages, the principal investigator will judge on a case-by-case basis whether regular use of certain medications will interfere with the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: AD group SPPA group HC group Partners
Sampling Method: Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Social Memory Test | 2 days
  Memory scores (from 0 to 10) on an experimental test (higher score means a better performance) in 3 different contexts of learning

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saliou P, Chavant J, Belliard S, Merck C, de La Sayette V, Wallon D, Martinaud O, Eustache F, Laisney M. MEM&SO protocol: understanding the determinants of social learning in neurodegenerative diseases. BMC Psychol. 2024 May 28;12(1):307. doi: 10.1186/s40359-024-01791-w. PMID 38807183